CLINICAL TRIAL: NCT04617873
Title: Deep Brain Stimulation and Spinal Cord Stimulation Therapy Improve Motor Function in Multiple System Atrophy With Predominant Parkinsonism: a Multi-center, Prospective, Open Label Clinical Trial
Brief Title: DBS and SCS Therapy Improve Motor Function in Multiple System Atrophy With Predominant Parkinsonism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: zhangyuqing (Other)
Responsible Party: Sponsor-Investigator, zhangyuqing, Clinical Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020005
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Multiple System Atrophy, Parkinson Variant (Disorder)
Keywords: Deep Brain Stimulation; Spine Cord Stimulation; Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep bain stimulation and Spinal cord stimulation therapy (Experimental): The patients in this group will receive bilateral STN-DBS and SCS stimulation
  Interventions: Procedure: Bilateral STN-DBS and T10-T12 SCS

INTERVENTIONS:
Procedure: Bilateral STN-DBS and T10-T12 SCS — simultaneous stimulation of bilaterally-STN-DBS combined with spinal cord stimulation

SUMMARY:
Multiple system atrophy (MSA) is a debilitating and fatal neurodegenerative disorder and symptomatic therapeutic strategies are still limited.The parkinsonian type of MSA (MSA-P) has parkinsonian symptoms as its prominent manifestation, although Deep brain stimulation (DBS) at the subthalamic nucleus or globus pallidus interna has been an established treatment for Parkinson's disease patients, it is mostly ineffective in MSA-P patients, the improvement in motor function as short-lasting and rapidly followed by the early appearance of freezing of gait (FOG) and postural instability that counteracted DBS benefits and often leads to significant disability and loss of quality of life. Recently, some pilot studies demonstrated the safety and significant therapeutic outcome of SCS for FOG.The purpose of this clinical study is to understand the effectiveness of DBS combined with SCS for symptomatic treatment of MSA-P.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a debilitating and fatal neurodegenerative disorder that characterized pathologically by α-synuclein (aSyn) accumulation in oligodendrocytes, the myelinating glial cells of the central nervous system (CNS), and symptomatic therapeutic strategies are still limited.

The parkinsonian type of multiple system atrophy (MSA-P) has parkinsonian symptoms as its prominent manifestation and may have an initial but short-lived response to levodopa (L-dopa). Deep brain stimulation (DBS) at the subthalamic nucleus (STN) or globus pallidus interna(GPi) has been an established treatment for Parkinson's disease(PD) patients with medically intractable fluctuations and has shown long-term efficacy to improve parkinsonian motor symptoms, such as bradykinesia, rigidity and rest tremor. However, DBS therapy is mostly ineffective in MSA patients. For the patients with MSA-P, improvement in motor function is short-lasting and rapidly followed by the early appearance of freezing of gait (FOG) and postural instability that counteracted DBS benefits and often leads to significant disability and loss of quality of life. Dopaminergic therapy or other symptomatic medications only offer limited alleviation of FOG and often lose their effect over time. Spinal cord stimulation (SCS) is a well-established therapy for treating chronic lower back or low limb pain neuropathic pain. Recently, some pilot studies demonstrated the safety and significant therapeutic outcome of SCS for FOG in PD, MSA-P and primary progressive freezing gait（PPFG）patients.

Can combined DBS with SCS be an alternative approach for symptomatic treatment of parkinsonian symptoms and gait-associated problems in patients with MSA-P? The purpose of this clinical study is to understand the combined treatment effectiveness for MSA-P.

It's a a multi-center, prospective, open label clinical study with a 12 months follow-up period. The intended study population is individuals suffering from multiple system atrophy with predominant parkinsonism. Each subject will complete an enrollment/screening/baseline visit, an DBS&SCS implant and activation visit, and 3 months, and 12months follow-up visits. Data collected at the enrollment visit after the consent process includes: demographics, baseline clinical status, MSA-related medical history, and inclusion/exclusion criteria assessment.Baseline assessment includes: Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III,New Freezing of Gait Questionnaire (NFOGQ), Gait and Fall Questionnaire (GFQ), PD-related quality of life (PDQ-39) and Berg Balance Scale(BBS). The participants will proceed to implantation after satisfying implant inclusion and exclusion criteria. Medtronic Model 3389 DBS electrodes (Medtronic, U.S.A.) will be implanted in the STN bilaterally using a stereotactic technique, connected to a dual-channel ACTIVA Neurostimulator (Medtronic); Paddle-shaped SCS electrode with 16 contacts (AdaptiveStim® 39, 565; Medtronic, USA) will be implanted into the epidural space at the thoracic levels ranging from T10 to T12. Electrode positions of DBS will be verified by postoperative CT-MRI image fusion and electrode position of SCS will be verified by X-ray. The stimulators will be turned on within 1 month after electrode implantation surgery. The stimulation parameters could vary freely, but medications will be kept constant during the study period. At the end of month 12, participants will enter the long-term follow-up in which medications could vary freely.

ELIGIBILITY:
inclusion criteria:

1. meet the clinical diagnostic criteria of possible MSA-P;
2. with moderate to severe parkinsonism motor symptoms;
3. accept levodopa treatment for at least 6 months, and stable medication dose for at least 4 weeks;

exclusion criteria:

1. severe orthostatic hypotension;
2. score of Hamilton Depression Scale is more than 24.
3. score of Mini-mental State Examination is less than 24;
4. elevated risks for bleeding
5. with evident lesions on MRI structural images at T8-12 spinal cord segment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
change in motor examination( Movement Disorders Society's revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III) at 3 months postoperatively | 3 months after surgery
  demonstrate the statistically significant difference in change of motor score (MDS-UPDRS III) from baseline( Off medication) to 3months(On stimulation/Off medication); MDS-UPDRS III ranges from 0 to 132, higher scores mean a worse outcome .
change in motor examination( Movement Disorders Society's revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III) at 12 months postoperatively | 12 months after surgery
  demonstrate statistically significant improvement in score of MDS-UPDRS III from Off stimulation/Off medication state to On stimulation/Off medication state at 12 months; MDS-UPDRS III ranges from 0 to 132, higher scores mean a worse outcome
change in PD-related quality of life(PDQ-39) | 12 months after surgery
  demonstrate statistically significant improvement in score of PDQ-39 from baseline to 12 months;PDQ-39 was used to evaluate the improvement in quality of life, ranged from 0 to 156, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
change in the score of Gait and Fall Questionnaire (GFQ) at 3 months postoperatively | 3 months after surgery
  demonstrate statistically significant improvement in score of GFQ from baseline to 3 months;GFQ range from 0 to 64, higher scores mean a worse outcome.
change in the score of Gait and Fall Questionnaire (GFQ) at 12 months postoperatively | 12 months after surgery
  demonstrate statistically significant improvement in score of GFQ from baseline to 12 months; GFQ ranges from 0 to 64, higher scores mean a worse outcome.
change in severity of freezing of gait (New Freezing of Gait Questionnaire,NFOGQ) at 3 months postoperatively | 3 months after surgery
  demonstrate statistically significant improvement in score of "New Freezing of Gait Questionnaire (NFOGQ)" from baseline to 3 months; NFOGQ is used to quantify freezing of gait severity, ranged from 0 to 30, higher scores mean a worse outcome.
change in severity of freezing of gait (New Freezing of Gait Questionnaire,NFOGQ) at 12 months postoperatively | 12 months after surgery
  demonstrate statistically significant improvement in score of "New Freezing of Gait Questionnaire (NFOGQ)" from baseline to 12 months; NFOGQ is used to quantify freezing of gait severity, ranged from 0 to 30, higher scores mean a worse outcome.
Clinical Global Impression-Global Improvement (CGI-GI) at 3 months postoperatively | 3 months after surgery
  to evaluate effectiveness on the basis of the physician's assessment, as well as on the basis of the patients' self-reported satisfaction. It is rated on a 7-point scale, range from 1(very much improved) through to 7 (very much worse)
Clinical Global Impression-Global Improvement (CGI-GI) at 12 months postoperatively | 12 months after surgery
  to evaluate effectiveness on the basis of the physician's assessment, as well as on the basis of the patients' self-reported satisfaction. It is rated on a 7-point scale, range from 1(very much improved) through to 7 (very much worse)
change in the score of Berg Balance Scale(BBS) at 3 months postoperatively | 3 months after surgery
  demonstrate statistically significant improvement in score of Berg Balance Scale(BBS) from baseline( Off medication state) to 3 months(On stimulation/Off medication state)； BBS ranged from 0 to 56, higher scores mean a better outcome.
change in the score of Berg Balance Scale(BBS) at 12 months postoperatively | 12 months after surgery
  demonstrate statistically significant improvement in score of Berg Balance Scale(BBS) from Off stimulation/Off medication state to On stimulation/Off medication state at 12 months；BBS ranged from 0 to 56, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Zhang, MD, Principal Investigator — Capital Medical University- Xuanwu Hospital
Locations (1):
- Capital Medical University of Xuanwu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No